CLINICAL TRIAL: NCT05774106
Title: The Therapeutic Relationship Between the Mental Health Case Manager and the Person With Severe Mental Health Disorder: a Mixed-methods Study
Brief Title: The Therapeutic Relationship Between the Case Manager and the Person With Severe Mental Health Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Instituto de Investigación Marqués de Valdecilla (Other); Col·legi Oficial Infermeres de Barcelona (Unknown)
Responsible Party: Principal Investigator, Marti Subias Miquel, Registered Mental Health Nurse, Principal Investigator, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PIC-60-22
Record Dates: First submitted 2022-12-21; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Mental Health Disorder; Case Management; Psychiatric Nursing
Keywords: action research; therapeutic relationship
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: First, a participatory intervention with nurses through the recording of four focus groups with the aim of understand, plan, change and maintain the practices surrounding the relationship therapy with their patients. Second, this intervention will be measured by administering scales to patients linked to the mental health case management program that provides service to different areas of the Barcelona Metropolitan Area. The variables to measure will be the quality of the therapeutic relationship, the recovery of the person and the overall functionality. These variables will be measured before and after finishing the participatory intervention.
Who Masked: Participant, Care Provider
Masking Description: A randomization of participating case managers will be performed. One intervention group will carry out the participatory action process and the other (control group) will carry out their professional activity normally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participatory Action Research (PAR). (Experimental): Two circular spirals following Kemmis & Mctaggart PAR principles. Each spiral includes the following stages: planning, action, observation and reflection.
  Four discussions groups and two reflective diaries will be carried out in total.
  Note: the PAR process will be conducted only with case managers.
  Interventions: Behavioral: Participatory action research
- Regular Practice (No Intervention): The other group will continue working as usual in their daily practice.

INTERVENTIONS:
Behavioral: Participatory action research — First, a participatory intervention with nurses through the recording of four focus groups with the aim of understand, plan, change and maintain the practices surrounding the relationship therapy with their patients. Second, this intervention will be measured by administering scales to patients linked to the mental health case management program that provides service to different areas of the Barcelona Metropolitan Area. The variables to measure will be the quality of the therapeutic relationship, the recovery of the person and the overall functionality. These variables will be measured before and after finishing the participatory intervention.
  Other Names: Critical Action Research
  Arms: Participatory Action Research (PAR).

SUMMARY:
The first mental health case management programs appear progressively in Spain from the trend towards community mental health with the aim of caring for people with severe mental health disorders outside from hospitals, accompanying them in their recovery process. The mental health nurse case manager is an example of advanced practice in in terms of assistance to the most seriously ill in the community mental health network.

The use of the therapeutic relationship as the central axis of care for the person is becomes an essential tool for patient recovery. This study aims, through participatory action, to inquire about the relationship therapy and its effect on the person's recovery. There will be a mixed methods research. First, a participatory intervention with nurses through the recording of four focus groups with the aim of understand, plan, change and maintain the practices surrounding the relationship therapy with their patients. Second, this intervention will be measured by administering scales to patients linked to the mental health case management program that provides service to different areas of the Barcelona Metropolitan Area. The variables to measure will be the quality of the therapeutic relationship, the recovery of the person and the overall functionality. These variables will be measured before and after finishing the participatory intervention. All data will be anonymized, transcribed and analyzed using the software correspondent.

DETAILED DESCRIPTION:
Two circular spirals following Kemmis & Mctaggart Participative Action Research (PAR) principles will be conducted. Each spiral includes the following stages: planning, action, observation and reflection.

Initially ( stage 0), the principal investigator will conduct an analysis of the current situation by observing, recording and analyzing the situation. The field diary will be used as a tool to assist in the data collection. Afterwards, a baseline measurement of the selected variables will be made by the principal investigator to both patients and participating professionals.

The first PAR cycle begins in January 2023: agreement and planning about how the observation of the therapeutic relationship will be carried out (focus group), the subsequent action-observation, which will be collected using a reflective diary, and the reflection in the discussion group based on the contributions of the reflective diaries, which will be contrasted with the available evidence with the aim of creating a dialogue.

The estimated duration of the first cycle is 2 months. The second cycle of PRA starts in March 2023: it begins with a focus group to discuss a new planning of strategies to implement changes. After a new period of action and self-observation of the changes (through reflective diary), the fourth and last group discussion group is held, with the purpose of sharing and evaluating the whole process. The estimated duration of this second cycle is 2 months.

At the end of the second cycle (May 2023), a follow-up measurement (post-test) will be carried out by the principal investigator. The estimated duration for this process is 1 month.

Note: the PAR process will be conducted only with case managers.

ELIGIBILITY:
Inclusion criteria of subjects

The following inclusion criteria have been pre-defined for professionals:

* Be a case management professional with one year of seniority in the program.
* To be available to carry out the PAR.

Regarding participating patients:

* To be treated at the Case management program (CMP). Have been diagnosed with a Severe Mental Health Disorder.
* No severe intellectual disability.
* Be between 18 and 65 years of age.
* Remain at the CMP during the 6-month duration of the intervention. Exclusion criteria for subjects. In reference to exclusion criteria, it is not contemplated to include case managers in the study who perform a substitution of less than 1 year's duration are not included in the study.

Similarly, exclusion from the study based on professional category is not contemplated.

Nor is it contemplated to include patients in whom the target intervention for which they were referred to the CMP program was the CMP program is less than 6 months (e.g., social emergencies, symptom control, psychoeducation at home, etc.),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-07-23 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify the meaning of the therapeutic relationship from the professional case manager's point of view. | 8 weeks
  It will be evaluated during the first cycle of the PAR, through the use of the discussion group (group reflection). All meetings will be recorded and coded using the Deddose platform for qualitative analysis.
Identify the meaning of the therapeutic relationship from the professional case manager's point of view. | 8 weeks
  It will be evaluated during the first cycle of the PAR, through the use of the reflective journal (individual self-analysis). All diaries will be transcribed and coded using the Deddose platform for qualitative analysis.
Determine strategies to improve the therapeutic relationship from the point of view of the professional case manager through reflection and discussion about evidence on therapeutic relationship avaliable | 8 weeks
  It will be evaluated during the second cycle of the PAR, through the use of the discussion group. All meetings will be recorded and coded using the Deddose platform for qualitative analysis.
Qualitatively evaluation of the implementation of improvement strategies in the therapeutic relationship | 4 weeks
  It will be evaluated at the end of the PAR's second cycle, through the use of the discussion group (group reflection) . All meetings will be recorded and coded using the Deddose platform for qualitative analysis.
Qualitatively evaluation of the implementation of improvement strategies in the therapeutic relationship | 4 weeks
  It will be evaluated at the end of the PAR's second cycle, through the use of the reflective journal (individual self-analysis). All diaries will be transcribed and coded using the Deddose platform for qualitative analysis.

SECONDARY OUTCOMES:
To identify the levels of prior therapeutic relationship between the professional case manager and the person with severe mental illness prior to the enhancement intervention in both the intervention and control groups. | 20 days
  A baseline measurement of the quality of the therapeutic relationship between the case manager and his or her patients prior to the beginning of the PAR will be carried out. "The Working Alliance Inventory - short" will be used. All data will be added to RedCap platform and analyzed with SPSS.
  *The Working Alliance Inventory-Short (WAI-S) is a refined measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. It's a 12 question scale with a list of of statements and questions about experiences people might have with their therapy or therapist. Each answers range from a Likert-type scale with five options: "seldom", "sometimes", "fairly often", "very often" and "always". The total score ranges from 12 to 84. The answer with the highest value depends on the statement of the phrase.
To identify the levels of prior therapeutic relationship between the professional case manager and the person with severe mental illness prior to the enhancement intervention in both the intervention and control groups. | 20 days
  A baseline measurement of the quality of the therapeutic relationship between the case manager and his or her patients prior to the beginning of the PAR will be carried out. The Quality of Psychiatric Care - Outpatient scale will be used. All data will be added to RedCap platform and analyzed with SPSS.
  *The QPC-OP consists of 30 items and measures six dimensions: Encounter (eight items), Participation (eight items), Discharge (four items), Support (four items), Secluded environment (three items), and Secure environment (three items). Each item begins with the sentence "I experience that..." and is assessed using a Likert-type scale with four options, going from 1 (totally disagree) to 4 (totally agree). The maximum score is 120 points and the minimum is 30 points. A high score in each dimension or for the scale as a whole indicates a perception of high quality both on the professional and it's patients.
To compare the results of the improvement intervention on the levels of therapeutic relationship with those previously identified. | 20 days
  When the intervention has been completed (PAR), a follow-up measurement will be taken using again "The Working Alliance Inventory - short version. All data will be added to RedCap platform and analyzed with SPSS.
  *The Working Alliance Inventory-Short (WAI-S) is a refined measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. It's a 12 question scale with a list of of statements and questions about experiences people might have with their therapy or therapist. Each answers range from a Likert-type scale with five options: "seldom", "sometimes", "fairly often", "very often" and "always". The total score ranges from 12 to 84. The answer with the highest value depends on the statement of the phrase.
To compare the results of the improvement intervention on the levels of therapeutic relationship with those previously identified. | 20 days
  When the intervention has been completed (PAR), a follow-up measurement will be taken using again "The The Quality of Psychiatric Care- Outpatient scale. All data will be added to RedCap platform and analyzed with SPSS.
  *The QPC-OP consists of 30 items and measures six dimensions: Encounter (eight items), Participation (eight items), Discharge (four items), Support (four items), Secluded environment (three items), and Secure environment (three items). Each item begins with the sentence "I experience that..." and is assessed using a Likert-type scale with four options, going from 1 (totally disagree) to 4 (totally agree). The maximum score is 120 points and the minimum is 30 points. A high score in each dimension or for the scale as a whole indicates a perception of high quality both on the professional and it's patients.
To compare the results with respect to levels of global functionality and perception of recovery at the end of the improvement intervention. | 8 weeks
  In addition to the quality of the therapeutic relationship, other variables will be measured. In the baseline and follow-up measurements, the patient's perception of recovery will also be measured, using the Recovery Assessment Scale.. All data will be added to RedCap platform and analyzed with SPSS.
  *The Recovery Assessment Scale (RAS) is a 20-item measure developed as an outcome measure for program evaluations. All items on the RAS assessment are rated on a 5-point Likert scale: 1 = Strongly Disagree, 2 = Disagree, 3 = Not Sure, 4 = Agree, and 5 = Strongly Agree. Responses are scored as a comprehensive total and as three separate domains: Clinical Recovery, Personal Recovery, and Social Recovery
To compare the results with respect to levels of global functionality and perception of recovery at the end of the improvement intervention. | 8 weeks
  In addition to the quality of the therapeutic relationship, other variables will be measured. In the baseline and follow-up measurements, the patient's functionality, using the "Health of the Nation Outcome Scale" scale. All data will be added to RedCap platform and analyzed with SPSS.
  *The Health of the Nation Outcome Scales (HoNOS) is a clinician rated instrument comprising 12 simple scales measuring behaviour, impairment, symptoms and social functioning for those in the 18 - 64 years old age group. Scores on each scale/item range from 0 (no problem) to 4 (severe problem).The total score ranging goes from 0 to 48 points.
To compare the results with respect to levels of global functionality and perception of recovery at the end of the improvement intervention. | 8 weeks
  In addition to the quality of the therapeutic relationship, other variables will be measured. In the baseline and follow-up measurements, the patient's functionality, using the "Camberwell Assessment of Need Short Appraisal Schedule" scale. All data will be added to RedCap platform and analyzed with SPSS.
  *The "Camberwell Assessment of Need Short Appraisal Schedule" scale assesses the health and social needs of adults across 22 domains of life, such as accommodation, food, self-care, daytime activities, psychotic symptoms, childcare, money, psychological distress, physical health and relationships. The need rating is made using the CAN rating algorithm: If the interviewee does not know or does not want to answer questions on this domain then rate ? (not known); If a current serious problem is present (regardless of cause, or whether any help is being given or not)then rate U (unmet need); If there is no serious problem because of help given then rate M (met need) otherwise Rate N

CONTACTS AND LOCATIONS:
Overall Officials: MARTI SUBIAS MIQUEL, Phd candidate, Principal Investigator — SJD Research Foundation
Locations (1):
- SJD Research Foundation, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No